CLINICAL TRIAL: NCT02558049
Title: Should I Continue Taking My Acid Reflux Medication? Development and Pilot Testing of a Patient Decision Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Wade Thompson, MSc student, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4393
Record Dates: First submitted 2015-09-17; First posted 2015-09-23 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Proton Pump Inhibitors; Gastroesophageal Reflux Disease
Keywords: Patient decision aid
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decision aid (Experimental): Patients will receive the patient decision aid during a 15 minute consultation with a clinical pharmacist.
  Interventions: Other: Decision aid

INTERVENTIONS:
Other: Decision aid — Participants will receive a patient decision aid which outlines the potential benefits and harms of proton pump inhibitor use, as well as the potential benefits and harms of switching to a lower dose of PPI or stopping and using on-demand (only when symptoms occur). The decision aid also allows participants to clarify their values regarding these potential benefits and harms.

SUMMARY:
BACKGROUND: Proton pump inhibitors (PPIs) treat problems such as gastroesophageal reflux disease (GERD). In many patients with mild or moderate GERD, PPIs should be used for 1-2 months but are often continued longer unnecessarily. This is a problem because PPIs may cause harm when used long-term. PPI use is associated with severe C. difficile infections, fractures and pneumonia. Canada's public drug programs spent $247 million on PPIs in 2012 (not including Quebec or PEI). Due to concerns with long-term PPI use, patients may face the decision to continue their PPI, use a lower dose or stop and use on-demand (only when symptoms return). This decision should be made collaboratively between patients and clinicians, though patients tend to have a poor understanding of when reducing a drug is appropriate. Using a lower dose or using on-demand may be viewed as difficult because of the chance of symptoms returning. Patient decision aids (PDAs) inform patients on benefits and risks of treatment options and improve ability to make informed decisions and clarify values. OBJECTIVES: Develop a PDA to help patients with the decision to continue PPI or stop and use on-demand/use a lower dose. Evaluate whether: 1) the PDA changes patient preference to continue or stop and use on-demand/use a lower dose of PPI 2) the PDA improves patient knowledge and realistic expectations 3) patients and pharmacists feel they made a shared decision 4) there is a change in PPI prescribing 8 weeks post-PDA and 5) patients' choices match up with their values. METHODOLOGY: The PDA will be developed by a team of doctors, pharmacists and patients. It will be delivered during a visit with a pharmacist. Patients (n=54) will indicate which choice they prefer (continue PPI/stop or use lower dose) before and after going through the PDA. We will use Mcnemar's test to compare the number of patients preferring to continue their PPI before and after. We will evaluate whether there is a difference in knowledge test scores and expectations test scores before and after the PDA. After the PDA, we will ask patients and pharmacists to rate the extent to which shared decision making occurred and measure the agreement. Values/choice congruence will be evaluated using logistic regression. Eight weeks after patients have received the PDA, we will look at whether there is any reduction in PPI use.

ELIGIBILITY:
Inclusion Criteria:

* Taking PPI for greater than or equal to 4 weeks, no current symptoms, taking PPI for mild to moderate upper GI symptoms (mild to moderate gastroesophageal reflux disease, grade A/B esophagitis)

Exclusion Criteria:

* Severe esophagitis (grade C/D), severe GERD or upper GI symptoms, currently experiencing upper GI symptoms, taking PPI for gastroprotection due to NSAID therapy (at moderate or high risk of GI bleed), history of Barrett's esophagus, history of bleeding peptic ulcer, taking PPI for treatment of current ulcer not healed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Decision preference (continue PPI or stop and use on-demand/use a lower dose) | Single visit - immediately before decision aid delivered (baseline), immediately after decision aid delivered (15 minutes)
  Difference in proportion of patients preferring to continue PPI therapy before and after PDA assessed using Mcnemar's test. The choice to continue will be the composite of patients wishing to continue and those unsure (since patients who are unsure would continue on PPI). We plan to conduct subgroup analysis based on decisional conflict at baseline for the primary outcome and secondary outcomes. Our subgroups will be (i) patients who are confident in their choice at baseline (SURE test score of 4) and (ii) patients who are not confident in their choice at baseline (SURE test score <4). The decision preference will be assessed at a single visit (before the PDA is delivered and right after).

SECONDARY OUTCOMES:
Change in Knowledge | Single visit - immediately before decision aid delivered (baseline), immediately after decision aid delivered (15 minutes)
  Difference in mean test score before and after assessed using paired t-test; two different versions of the knowledge test will be used
Change in Realistic expectations | Single visit - immediately before decision aid delivered (baseline), immediately after decision aid delivered (15 minutes)
  Difference in mean test score before and after assessed using paired t-test
Values/choice congruence | Single visit - after decision aid is delivered (15 minutes)
  Multiple logistic regression with dichotomous outcome of continue PPI or stop/use a lower dose of PPI and the following variables: value rating (continuous measure from 1-5, 1: favours deprescribing - 5: favours continuation), age, gender, level of education. Conducted in patients passing knowledge test (>50% score).
Agreement in rating of extent of shared decision-making | Single visit - immediately after decision aid is delivered (15 minutes)
  Agreement between pharmacist and participant rating measured using kappa coefficient
Change in Decisional conflict (SURE test) | Single visit - immediately before decision aid delivered (baseline), immediately after decision aid delivered (15 minutes)
  Paired t test comparing SURE score before and after patient receives PDA
Change in PPI prescription | 8 weeks after decision aid is delivered
  95% confidence interval around the proportion of patients whose PPI prescription is changed after 8 weeks
Clinical symptoms at 8 weeks | 8 weeks after decision aid is delivered
  Compare the proportion of patients whose symptoms have returned for patients who continued their PPI versus those who switched to a lower dose or stopped and used on-demand

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Elisabeth Bruyere Hospital, Ottawa, Ontario
  - Melrose FHT, Ottawa, Ontario
  - Rideau FHT, Ottawa, Ontario

REFERENCES:
- [Background] Katz PO, Gerson LB, Vela MF. Guidelines for the diagnosis and management of gastroesophageal reflux disease. Am J Gastroenterol. 2013 Mar;108(3):308-28; quiz 329. doi: 10.1038/ajg.2012.444. Epub 2013 Feb 19. No abstract available. PMID 23419381
- [Background] Ramakrishnan K, Salinas RC. Peptic ulcer disease. Am Fam Physician. 2007 Oct 1;76(7):1005-12. PMID 17956071
- [Background] Leri F, Ayzenberg M, Voyce SJ, Klein A, Hartz L, Smego RA Jr. Four-year trends of inappropriate proton pump inhibitor use after hospital discharge. South Med J. 2013 Apr;106(4):270-3. doi: 10.1097/SMJ.0b013e31828db01f. PMID 23558416
- [Background] Kwok CS, Arthur AK, Anibueze CI, Singh S, Cavallazzi R, Loke YK. Risk of Clostridium difficile infection with acid suppressing drugs and antibiotics: meta-analysis. Am J Gastroenterol. 2012 Jul;107(7):1011-9. doi: 10.1038/ajg.2012.108. Epub 2012 Apr 24. PMID 22525304
- [Background] Yu EW, Bauer SR, Bain PA, Bauer DC. Proton pump inhibitors and risk of fractures: a meta-analysis of 11 international studies. Am J Med. 2011 Jun;124(6):519-26. doi: 10.1016/j.amjmed.2011.01.007. PMID 21605729
- [Background] Spijker-Huiges A, Winters JC, Meyboom-De Jong B. Patients' views on dyspepsia and acid suppressant drug therapy in general practice. Eur J Gen Pract. 2006;12(1):10-4. doi: 10.1080/13814780600757120. PMID 16945866
- [Background] Reeve E, To J, Hendrix I, Shakib S, Roberts MS, Wiese MD. Patient barriers to and enablers of deprescribing: a systematic review. Drugs Aging. 2013 Oct;30(10):793-807. doi: 10.1007/s40266-013-0106-8. PMID 23912674
- [Background] Coulter A, Stilwell D, Kryworuchko J, Mullen PD, Ng CJ, van der Weijden T. A systematic development process for patient decision aids. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S2. doi: 10.1186/1472-6947-13-S2-S2. Epub 2013 Nov 29. PMID 24625093
- [Background] Durand MA, Witt J, Joseph-Williams N, Newcombe RG, Politi MC, Sivell S, Elwyn G. Minimum standards for the certification of patient decision support interventions: feasibility and application. Patient Educ Couns. 2015 Apr;98(4):462-8. doi: 10.1016/j.pec.2014.12.009. Epub 2014 Dec 31. PMID 25577469
- [Background] Legare F, Turcotte S, Stacey D, Ratte S, Kryworuchko J, Graham ID. Patients' perceptions of sharing in decisions: a systematic review of interventions to enhance shared decision making in routine clinical practice. Patient. 2012;5(1):1-19. doi: 10.2165/11592180-000000000-00000. PMID 22276987
- [Background] Lachenbruch PA. On the sample size for studies based upon McNemar's test. Stat Med. 1992 Aug;11(11):1521-5. doi: 10.1002/sim.4780111110. PMID 1410964
- [Background] Janz NK, Wren PA, Copeland LA, Lowery JC, Goldfarb SL, Wilkins EG. Patient-physician concordance: preferences, perceptions, and factors influencing the breast cancer surgical decision. J Clin Oncol. 2004 Aug 1;22(15):3091-8. doi: 10.1200/JCO.2004.09.069. PMID 15284259
- See also: Decision Aid Toolkit — https://decisionaid.ohri.ca/resources.html